CLINICAL TRIAL: NCT04555018
Title: Correlation Between Dehydroepiandrosterone Sulfate and Sebum Level in Adult Female Acne Vulgaris
Status: Completed | Type: Observational
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Irma Bernadette S. Sitohang, MD, PhD - Head of Division of Cosmetic Dermatology, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Organization: Indonesia University (Other)
Other Study IDs: DheasSebum
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Acne Vulgaris; Female
Keywords: Acne vulgaris; Sebum level; Dehydroepiandrosterone Sulfate
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the correlation between Dehydroepiandrosterone sulfate (DHEAS) and sebum level in adult female acne. A cross sectional study was conducted with 50 samples, in June to October 2017.

DETAILED DESCRIPTION:
Epidemiological studies have shown that number of adult female acne vulgaris (AV) increases. Hormone, sebum production, Propionibacterium acne and inflammatory process are factors involved in AV development. The aim of this study is to determine the correlation between Dehydroepiandrosterone sulfate (DHEAS) and sebum level in adult female acne. This research used cross sectional study with 50 samples, aged 25-49 years by consecutive sampling. The degree of acne vulgaris was evaluated using Lehman criteria , and then the sebum level and DHEAS were measured objectively using sebumeter and serum, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 25-29 years
* Diagnosed with mild to severe acne vulgaris
* Agree to participate

Exclusion Criteria:

* History of taking antiandrogen drugs
* History of taking oral and topical antibiotics, using topical retinoid and BPO in the last 4 weeks
* History of taking oral isotretinoin in the last 6 months
* Pregnancy or breastfeeding

Ages: 25 Years to 49 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Female , age 25-29 years, diagnosed with mild to severe acne vulgaris
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Sebum level | One day
  Using sebumeter to evaluate the sebum level objectively
Dehydroepiandrosterone sulfate | One day
  Blood serum was used to evaluate Dehydroepiandrosterone sulfate level.

CONTACTS AND LOCATIONS:
Overall Officials: Irma B Sitohang, MD,PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Indonesia dr. Cipto Mangunkusumo Hospital, Jakarta, Jakarta Pusat, Indonesia